CLINICAL TRIAL: NCT01663922
Title: Phase I Evaluation of the Pharmacokinetics and Safety of Boceprevir and Ucalm (St John&Apos;s Wort) When Co-administered to Male and Female Healthy Volunteers.
Brief Title: Boceprevir and Ucalm (St John&Apos;s Wort)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: University of Liverpool (Other); University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SSAT 045
Record Dates: First submitted 2012-08-03; First posted 2012-08-13 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Hypericum extract LI 160; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- St John's Wort, then Boceprevir (Experimental): D 1-14 St. John's Wort 2 x 300mg (Ucalm(r)) QD D 22-35 St. John's Wort 2 x 300mg (Ucalm(r)) QD D 31-35 Boceprevir 800mg tds D 52-56 Boceprevir 800mg tds
  Interventions: Drug: Boceprevir; Drug: St John's Wort
- Boceprevir, then St John's Wort (Experimental): D 10-14 Boceprevir 800mg tds D 22-35 St. John's Wort 2 x 300mg (Ucalm(r)) QD D 31-35 Boceprevir 800mg tds D 43-56 St. John's Wort 2 x 300mg (Ucalm(r)) QD
  Interventions: Drug: Boceprevir; Drug: St John's Wort

INTERVENTIONS:
Drug: Boceprevir — Boceprevir as Victrelis(r) 200mg capsules
  Other Names: Boceprevir 800 mg three times daily
Drug: St John's Wort — Each Ucalm(r) tablet contains 300mg of St Johns Wort extract
  Other Names: Ucalm (R) tablets, two tablets given once daily

SUMMARY:
The purpose of the study is to look at whether taking a new medication for hepatitis C (boceprevir) together with a herbal remedy commonly used for the treatment of depression (SJW) has any effect on the levels of boceprevir in the blood, compared to when boceprevir is taken on its own.

Treatment of hepatitis C genotype-1, has recently been significantly improved with the addition of a new class of drugs called protease inhibitors (PIs). Boceprevir belongs to this class of antiviral drugs and it is administered in combinations with other drugs to treat hepatitis C. One of the common side effects of treatment for hepatitis C is low mood (depression) for which treated patients may self-medicate with preparations containing St. Johns Wort (SJW).

SJW is known to cause drug interactions, so taking SJW at the same time as boceprevir may result in a change in how both of these drugs usually work. It is therefore important to find out if the levels of boceprevir in the blood are significantly affected by taking SJW.

The study aims to help us understand whether it will be safe to take SJW whilst being simultaneously treated for hepatitis C with boceprevir.

DETAILED DESCRIPTION:
Boceprevir is a strong inhibitor of CYP3A4/5. Medicines metabolized primarily by CYP3A4/5 may have increased exposure when administered with boceprevir, which could increase or prolong their therapeutic and adverse reactions. Boceprevir does not inhibit or induce the other enzymes of the CYP450 family.

Boceprevir has been shown to be a P-glycoprotein and breast cancer resistant protein (BCRP) substrate in vitro. There is potential for inhibitors or inducers of these transporters to alter the concentrations of boceprevir; the clinical implications of these interactions are not known.Boceprevir is partly metabolized by CYP3A4/5. Co-administration of boceprevir with medicines that induce or inhibit CYP3A4/5 could increase or decrease exposure to boceprevir and affect its efficacy.Boceprevir, in combination with peginterferon and ribavirin, is contraindicated when coadministered with medicines that are highly dependent on CYP3A4/5 for clearance, and for which elevated plasma concentrations are associated with serious and/or life-threatening events. Examples may include; orally administered midazolam and triazolam, bepridil, pimozide, lumefantrine, halofantrine, and tyrosine kinase inhibitors, and ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine).

Boceprevir is primarily metabolized by aldoketo reductase (AKR). In medicine interaction trials conducted with AKR inhibitors diflunisal and ibuprofen, boceprevir exposure did not increase to a clinically significant extent. Boceprevir may be co-administered with AKR inhibitors. The concomitant use of boceprevir with stong CYP3A4 inducers such as rifampicin or anticonvulsants (such as phenytoin, phenobarbital or carbamazepine) may significantly reduce the plasma exposure of boceprevir. As no data is available, the combination of boceprevir with these medicines is not recommended.

The metabolism of St John's Wort is not currently known. Treatment with St John's wort for 14 days resulted in significant increases in the urinary 6-beta-hydroxycortisol/ cortisol ratio, suggesting that St John's wort is an inducer of CYP3A4. For this reason, it is not recommended to administer SJW with CYP3A4 metabolized drugs. Furthermore,interactions may occur with P-glycoprotein substrates, as St. John's wort can induce the activity of transmembrane transporters. This might decrease the effectiveness of some medications.

For the reasons illustrated above, the potential for a drug interaction between SJW and boceprevir is high and the co-administration must be studied in order to gain information on whether: i) SJW leads to a decrease in boceprevir concentrations and therefore efficacy; ii) boceprevir leads to an increase in SJW (hypericin) exposure with risk of toxicity.

The safety and PK of the combination should be known especially in view of the common side effects caused by interferon, which is co-administered with boceprevir for the treatment of hepatitis C: as interferon causes depression, patients may chose to take SJW rather than prescribed anti-depressants to manage their mood changes during antihepatitis treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 28 days prior to day 0:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
5. Women of childbearing potential (WOCBP), who are sexually active, must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least one month after the study in addition to the consistent and correct use of a condom. Examples of adequate methods of contraception for females in this trial are diaphragm with spermicide, substance and intra-uterine device. Hormonal contraceptives should not be considered a method of contraception and should be avoided if containing drospirenone.
6. Willing to consent to their personal details being entered onto The Over volunteering Prevention Scheme (TOPS) database.
7. Registered with a GP in the UK
8. Willing to bring photo ID to each visit

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B and/or C antibodies
4. Positive blood screen for HIV-1 and 2 antibodies
5. Current or recent (within three months) gastrointestinal disease
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
7. Exposure to any investigational drug or placebo within three months of first dose of study drug (additional check to be made on TOPS www.tops.org.uk).
8. Consumption of grapefruit or Seville oranges, or any grapefruit or Seville orange containing product within one week of first dose of study drug and for the duration of the study
9. Use of any other drugs, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs (note OCPs containing drosperinone should be excluded)
10. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 30 days after the end of the treatment period
11. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — HIV Consultant
Locations (1):
- St Stephen's AIDS Trust, London, United Kingdom

REFERENCES:
- [Result] Jackson A, D'Avolio A, Moyle G, Bonora S, Di Perri G, Else L, Simiele M, Singh GJ, Back D, Boffito M. Pharmacokinetics of the co-administration of boceprevir and St John's wort to male and female healthy volunteers. J Antimicrob Chemother. 2014 Jul;69(7):1911-5. doi: 10.1093/jac/dku060. Epub 2014 Mar 6. PMID 24610312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All volunteers were recruited at a single centre, SSAT Research Unit, Chelsea & Westminster Hospital, London, UK.
Pre-assignment Details: Eligible participants took:
  SJW for 14 days Group A D1-D14 or boceprevir(BCP) for 5 D10-D14 days Group B (D 10-14); PK profile on D14 then 7 day washout period to D21 D22-D35, all took SJW (+ BCP on D31-D35); PK on D35 then washout to D42 Group A took BCP on D52-D56; Group B SJW on D43-D56; PK profile on D56.
Groups:
- Group A (St John's Wort Then Boceprevir): * St John's Wort, (SJW) for 14 days (1-14)
  * [wash out for 7 days (15-21)]
  * SJW for 14 days (22-35) plus boceprevir from day 31 to day 35 (5 days in total)
  * [wash out for 7 days (36-42)]
  * boceprevir from day 52 to day 56
- Group B (Boceprevir Then St John's Wort): * Boceprevir for 5 days (10-14)
  * [wash out for 7 days (15-21)]
  * SJW for 14 days (22-35) plus boceprevir from day 31 to day 35 (5 days in total)
  * [wash out for 7 days (36-42)
  * SJW from day 43 to day 56
Period: First Intervention (14 Days or 5 Days)
Arm/Group | Group A (St John's Wort Then Boceprevir) | Group B (Boceprevir Then St John's Wort)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Group A (St John's Wort Then Boceprevir) | Group B (Boceprevir Then St John's Wort)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Group A (St John's Wort Then Boceprevir) | Group B (Boceprevir Then St John's Wort)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Group A (St John's Wort Then Boceprevir) | Group B (Boceprevir Then St John's Wort)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Third Intervention (14 Days or 5 Days)
Arm/Group | Group A (St John's Wort Then Boceprevir) | Group B (Boceprevir Then St John's Wort)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Participants: Descriptive analysis of combined groups
Arm/Group | All Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic of Boceprevir in the Presence of Ucalm (St John's Wort)
Description: Pharmacokinetic parameters (maximum and trough concentrations, and area under concentratof boceprevir and SJW will be evaluated when given in combination at steady-state to evaluate possible differences in concentrations during co-administration versus drug given alone.
  The pharmacokinetic parameters calculated for boceprevir and SJW will be Ctrough,the maximum observed plasma concentration (Cmax), time point at Cmax (Tmax), and total drug exposure, expressed as the area under the plasma concentration-time curve.
  All pharmacokinetic parameters will be calculated using non-compartmental modelling techniques (WinNonlin®) and all statistical calculations performed within-participant changes in the assessed pharmacokinetic parameters (drug alone vs drug combination) will be evaluated by calculating geometric mean ratios.
Time Frame: 6 months
Population: All participants who completed the three PK assessments were included in the analysis. BCP metabolites (SCH534128 & SCH523129) PK parameters were determined in the presence and absence of SJW, and hypericin PK parameters in the presence and absence of BCP; for the total study population.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Groups:
- All Participants: Combined analysis of both group sequences
Arm/Group | All Participants
Number analyzed (Participants) | 17
ng*h/mL
  Total Boceprevir alone | 4588 [4160 to 5317]
  Boceprevir in presence of St Johns Wort) | 4204 [3785 to 4886]
  Hypericin alone | 11.6 [9.3 to 17.0]
  Hypericin in presence of boceprevir | 14.3 [11.2 to 20.8]
  SCH534128 alone | 3222 [2929 to 3687]
  SCH534128 in presence of St. Johns Wort | 2935 [2653 to 3687]

ADVERSE EVENTS:
Groups:
- Group A: St John's Wort first
- Group B: Boceprevir first
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 6/8 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=8) | Group B (N=9)
Headache (Nervous system disorders) | 4 (5) | 3 (9)
coryzal symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (7)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
nausea (Nervous system disorders) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
pre-syncope (Cardiac disorders) | 0 (0) | 1 (1)
dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
conjunctival infection (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No